CLINICAL TRIAL: NCT04531449
Title: An Observational Study to Determine the Usability of the Inflammacheck Device by Healthcare Providers in the Intended Use Environment - EXhaled Hydrogen Peroxide As a Marker of Lung diseasE Study - Conformité Européenne
Brief Title: EXhaled Hydrogen Peroxide As a Marker of Lung Disease Study - Conformité Européenne (European Conformity)
Acronym: EXHALE CE
Status: Completed | Type: Observational
Sponsor: Portsmouth Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: PHT/2019/44
Record Dates: First submitted 2020-08-21; First posted 2020-08-28 (Actual); Last update posted 2020-08-28 (Actual); Status verified 2020-08

CONDITIONS: Point of Care Monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is designed to test whether the Inflammacheck™ device is easy to use by healthcare professionals who would be using it in a clinic setting or in primary care. The data collected during this study will be used as part of the evidence needed to get the CE (Conformité Européenne) marking for the device.

CE marking is a certification mark that indicates conformity with health, safety, and environmental protection standards for products sold within the European Economic Area (EEA). CE marking is essential for any medical devices used in the UK or the EU.

DETAILED DESCRIPTION:
This observational study has been designed to evaluate the ability of healthcare providers to use the Inflammacheck™, an investigational medical device, to measure participants exhaled breath condensate (EBC) H2O2. The data will be used to support the CE marking of the Inflammacheck™ device.

A measure of the participants' EBC H2O2 will be measured on the Inflammacheck™ device to demonstrate usability and comprehension of the instructions for use.

There are no control measurements involved in the study, all of the participants' EBC H2O2 measurements will be performed using Inflammacheck™ only.

Only healthcare providers naïve to the Inflammacheck™ device will be eligible to take part in the assessment of usability. This is to ensure that the usability assessment will not be biased by prior knowledge of the device or its instructions. The only training provided will be an introductory presentation explaining the Clinical Investigation objectives.

The total time for participant involvement is one session comprising of:

* Information & consent
* EBC H2O2 measurement with Inflammacheck™

ELIGIBILITY:
Inclusion Criteria:

* Male or Female, aged 18 years or above.
* Member of NHS staff at PHT.
* Is a healthcare provider.
* Participant is willing and able to give informed consent for participation in the study.

Exclusion Criteria:

* In the opinion of the clinical investigator, participant could be put at risk of harm by having to perform any of the study procedures.
* Unable to comprehend the study and provide informed consent e.g. insufficient command of English in the absence of someone to adequately interpret.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: NHS staff
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2019-06-06 (Actual); Primary Completion 2019-10-09 (Actual); Study Completion 2019-10-09 (Actual)

PRIMARY OUTCOMES:
To determine the usability of the Inflammacheck device in health care providers | immediately after the procedure
  number of attempts taken to obtain a result

CONTACTS AND LOCATIONS:
Locations (1):
- Portsmouth Hospitals NHS Trust, Queen Alexandra Hospital, Portsmouth, Hampshire, United Kingdom